CLINICAL TRIAL: NCT04208139
Title: A Random Selection of Patients From the SENTRY Study Who Have a Bioconverted Sentry IVC Filter in Situ With a Minimum Dwell Time of 24 Months From a Single Center
Brief Title: A Random Selection of Patients From the SENTRY Study Who Have a Bioconverted Sentry IVC Filter in Situ With a Minimum Dwell Time of 24 Months From a Single Center Follow up
Status: Completed | Type: Observational
Sponsor: NC Heart and Vascular Research, LLC (Other)
Collaborators: Novate Medical Limited, a BTG Group Company (Unknown)
Responsible Party: Sponsor
Other Study IDs: Version 1.0
Record Dates: First submitted 2019-12-03; First posted 2019-12-23 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2019-12

CONDITIONS: Recurrent Pulmonary Embolism (Disorder)
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Diagnostic Test: IVUS — IVUS

SUMMARY:
IVUS Evaluation of the Bioabsorbable Sentry IVC Filter 3-5 Years Post Deployment Follow up

DETAILED DESCRIPTION:
IVUS Evaluation of the Bioabsorbable Sentry IVC Filter 3-5 Years Post Deployment Follow up

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Signed the informed consent document
* Participants from the SENTRY clinical trial willing to undergo one time IVUS evaluation ( outpatient )

Exclusion Criteria:

* Any filter that remained non converted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with at least 24 months dwell time will undergo IVUS assessment of the inferior vena cava
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2020-03-14 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Patency of the inferior vena cava | 3-5 years
Cylindrical frame integrity | 3-5 years
  Cylindrical frame integrity
Impact of the Sentry cylindrical frame on the vessel wall evaluation for endothelialization and neointimal hyperplasia and wall dynamics | 3-5 years
  Impact of the Sentry cylindrical frame on the vessel wall evaluation for endothelialization and neointimal hyperplasia and wall dynamics
Presence and characterization of adherent thrombus | 3-5 years
  Presence and characterization of adherent thrombus

CONTACTS AND LOCATIONS:
Locations (1):
- NC Heart and Vascular Research, LLC, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No